CLINICAL TRIAL: NCT05243420
Title: Commonly Used Drug Regimens for Rapid Sequence Intubation (RSI) of Trauma Patients in the Emergency Department
Status: Withdrawn | Type: Observational
Why Stopped: Unable to obtain IRB approval and data agreements prior to request for data submission. No subjects were enrolled and no study activities have occurred.
Sponsor: Methodist Health System (Other)
Collaborators: University of Texas at Austin (Other)
Responsible Party: Sponsor
Other Study IDs: 069.GME.2019.D
Record Dates: First submitted 2020-09-22; First posted 2022-02-17 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Trauma Patients

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Airway is the first step in the initial assessment of a trauma patient. Often this assessment determines the need for endotracheal intubation, most commonly by rapid sequence intubation (RSI). Currently, there is no consensus on best practice for RSI drug regimens. Given the fragmented nature of this topic, most RSI drugs are chosen by the intubating physician based on their experience (i.e., a "dealer's choice"). Overall, emergency medical care is moving towards standardization to decrease medical errors and improve outcomes. Clearly, the current approach to RSI drug regimens does not align with those goals.

This study seeks first to define commonly used RSI drug regimens for trauma, and second to investigate hospital course and long-term health outcomes as a potential way to define best practice RSI drugs for trauma patients.

The study will be a multi-center retrospective chart review of data collected from January 1, 2014 to January 1, 2019, and will include Level I trauma centers in Texas. The University of Texas at Austin (UTA) is hosting this study as a Texas Level I Trauma Centers Multicenter Trial. Additional sites will have their own institutional IRB approval and will provide de-identified data to the principal investigator (PI) via secure encrypted email. Data will be submitted for MDMC trauma patients to UTA and analyzed within the Dell Med Department of Surgery and Perioperative Care and treated in the same way with the same security as data collected at Dell Seton Medical Center. The plan to complete the data collection and analysis by January 1, 2021.

After de-identification, descriptive statistical analysis will be performed. Statistics reported will include frequencies. Logistic regression model to predict outcome will be performed. Odds ratio, confidence interval, and P value will be reported using logistic regression for outcome models for both adjusted and unadjusted models. The statistical software package SAS 9.3 will be used for all calculations.

DETAILED DESCRIPTION:
Airway is the first step in the initial assessment of a trauma patient. Often this assessment determines the need for endotracheal intubation, most commonly by rapid sequence intubation (RSI). Currently, there is no consensus on best practice for RSI drug regimens. The research on drugs for RSI mainly focused on immediate hemodynamic effect, number of intubation attempts, and, more recently, adrenal insufficiency related to etomidate administration. There is little research, and no American multicenter research, on non-immediate health outcomes such as mortality. Additionally, there is a growing body of literature that suggests trauma patients may respond differently to RSI regimens than other critically ill patients. Given the fragmented nature of this topic, most RSI drugs are chosen by the intubating physician based on their experience (i.e., a "dealer's choice"). Overall, emergency medical care is moving towards standardization to decrease medical errors and improve outcomes. Clearly, the current approach to RSI drug regimens does not align with those goals.

There are three major gaps in the literature. First, there is no definition of the commonly used RSI drug regimens for trauma patients. It is essential to define common RSI drug regimens in order to facilitate future research and analyze drug efficacy. Second, the unique response of trauma patients to RSI drugs has not been elucidated. Third, there is little description of short and long term (vs. solely short term) outcomes for each of the RSI regimens. This will be an essential piece of information when discussing standardization and deciding which regimens are best suited for patients.

This study seeks first to define commonly used RSI drug regimens for trauma, and second to investigate hospital course and long-term health outcomes as a potential way to define best practice RSI drugs for trauma patients.

The study will be a multi-center retrospective chart review of data collected from January 1, 2014 to January 1, 2019, and will include Level I trauma centers in Texas. The University of Texas at Austin (UTA) is hosting this study as a Texas Level I Trauma Centers Multicenter Trial. Additional sites will have their own institutional IRB approval and will provide de-identified data to the principal investigator (PI) via secure encrypted email. Data will be submitted for MDMC trauma patients to UTA and analyzed within the Dell Med Department of Surgery and Perioperative Care and treated in the same way with the same security as data collected at Dell Seton Medical Center. After data abstraction, the PI will de-identify data before analysis, removing name, and medical record number (MRN). All data recording and collection will include a computer, which is secured via password. Documents will be password protected, hosted on UT Box, and only downloaded after de-identification. Only the PI, Co-PI, and research coordinators will have access to the data. The dataset will be password protected. No identifiable health information will be used in reporting of data, whether that is in publication or presentation format. The investigators plan to complete the data collection and analysis by January 1, 2021.

After de-identification, descriptive statistical analysis will be performed. Statistics reported will include frequencies. Logistic regression model to predict outcome will be performed. Odds ratio, confidence interval, and P value will be reported using logistic regression for outcome models for both adjusted and unadjusted models. The statistical software package SAS 9.3 will be used for all calculations.

ELIGIBILITY:
Inclusion Criteria:

* Any adult (18 to 89 years old)
* Traumatic injury
* Intubation attempt made in the emergency department

Exclusion Criteria:

* Prisoners
* Pregnant Women
* Patients less than 18 years of age

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult trauma patients with intubation attempt in emergency department
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Commonly Used Drug Regimens for Rapid Sequence Intubation (RSI) of Trauma Patients in the Emergency Department | January 1, 2014 to January 1, 2019
  Commonly Used Drug Regimens for Rapid Sequence Intubation (RSI) of Trauma Patients in the Emergency Department
Demographics | January 1, 2014 to January 1, 2019
  Age (in years)
Prehospital vitals | January 1, 2014 to January 1, 2019
  Vital signs collected prior to hospitalization
Emergency department vitals | January 1, 2014 to January 1, 2019
  Vitals recorded in the emergency department
Peri-intubation vitals | January 1, 2014 to January 1, 2019
  Vitals recorded prior to intubation
AIS | January 1, 2014 to January 1, 2019
  (Abbreviated Injury Score)
Death Rate | January 1, 2014 to January 1, 2019
  rate of death
ISS | January 1, 2014 to January 1, 2019
  (Injury Severity Score)
Hospital Length of Stay | January 1, 2014 to January 1, 2019
  The number of days subject was admitted.
ICU Length of Stay | January 1, 2014 to January 1, 2019
  The number of days the subject was admitted into the ICU.
Ventilation days | January 1, 2014 to January 1, 2019
  The number of days the subject ventilated.
Return to Hospital in <30d | January 1, 2014 to January 1, 2019
Discharge Disposition | January 1, 2014 to January 1, 2019
  discharge status
Demographics-Sex | January 1, 2014 to January 1, 2019
  Male or female
Demographics-Race | January 1, 2014 to January 1, 2019
  Race of subject
Demographics-Trauma Type | January 1, 2014 to January 1, 2019
  Type of trauma

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Truitt, MD, Principal Investigator — Methodist Health System
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No